CLINICAL TRIAL: NCT01218412
Title: Investigation of Web-based Motivational Interviewing to Increase Physical Activity Participation Among Adults
Brief Title: Web-based Physical Activity Program
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karnes, Sasha (Individual)
Collaborators: University of Wisconsin, Whitewater (Other)
Responsible Party: Principal Investigator, Sasha Karnes, Ph.D., Karnes, Sasha
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 10-84E
Record Dates: First submitted 2010-10-04; First posted 2010-10-11 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2014-04

CONDITIONS: Physical Activity
Keywords: Physical Activity; Motivational Interviewing; Web-based; Physician Referral
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Web-based, Mi=Based Intervention (Experimental): 4 session web-based, MI-based intervention.
  Interventions: Behavioral: Web-based Motivational Interviewing

INTERVENTIONS:
Behavioral: Web-based Motivational Interviewing — Participants will engage in 4 sessions of web-based motivational interviewing over the course of 4 weeks.

SUMMARY:
The specific aims of the proposed study are:

* 1. To determine if web-based Motivational Interviewing (MI) is effective, compared to an informational web-based comparison group, in enhancing physical activity (PA) participation; and
* 2. To assess the mechanisms by which web-based MI enhances PA through changes in targeted cognitive mediators.

The specific hypotheses of the study include that:

* Hypothesis 1: Web-based MI will increase PA;
* Hypothesis 2: Web-based MI will lead to stage progression in the direction of increased readiness to participate in PA;
* Hypothesis 3: Web-based MI will influence theoretically identified cognitive variables;
* Hypothesis 4: Cognitive variables will mediate increases in PA participation.

DETAILED DESCRIPTION:
Increasing physical activity (PA) is a public health priority. There is preliminary support for application of Motivational Interviewing (MI) for physical activity (PA), web-applications for PA promotion, web-based MI for behavior change, and finally web-based MI for PA. Based on collective findings in these areas of inquiry, it is necessary to investigate the efficacy of MI as a method that lends readily to practical applications for PA promotion. The current study seeks to investigate whether web-based MI can be applied in an adult population to enhance PA participation using a physician referral scheme. Additionally, mechanisms of behavior change are considered in order to inform future research and intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults referred through primary care due to insufficient physical activity standards based on Centers for Disease Control (CDC) guidelines for aerobic activity.
* Must have internet access and e-mail.
* Cleared by physician for physical activity participation.

Exclusion Criteria:

* Greater than 10,000 steps per day on average based on baseline pedometer screening over the course of 7 days.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 132 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Physical Activity (pedometer recordings) | 1 week post-intervention
  Physical activity will be assessed using pedometers.
Physical activity (self-report) | 3-months post-intervention
  Physical activity will be assessed using a self-report inventory.

SECONDARY OUTCOMES:
Cognitive Mediators | 3 months post intervention
  Cognitive mediators of physical activity participation including self-efficacy, readiness to change, motivation, intention, enjoyment, and decisional balance for physical activity will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Sasha L. Karnes, M.S., Principal Investigator — University of Wisconsin, Milwaukee
Locations (1):
- Aurora RiverCenter, Milwaukee, Wisconsin, United States